CLINICAL TRIAL: NCT04368741
Title: Effectiveness and Safety of Nutrition Product in Gestational Diabetes Mellitus Patients, Based on Continuous Glucose Monitoring, a Prospective Randomized Controlled Trial
Brief Title: Nutrition Product Combine With Continuous Glucose Monitoring in Gestational Diabetes Mellitus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: San MediTech(Huzhou)Co.,Ltd. (Unknown); Sanz Pharmaceutical Group (Unknown); Beijing Chao Yang Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ZS-2103
Record Dates: First submitted 2019-12-01; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-08

CONDITIONS: SANZ®KINGWILL Combined With CGM Equipment in GDM Patients; GLUCERNA SR® Combined With CGM Equipment in GDM Patients
Keywords: nutrition product; continuous glucose monitoring; gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucerna

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): SANZ®KINGWILL
  Interventions: Dietary Supplement: SANZ®KINGWILL
- Control group (Other): GLUCERNA SR®
  Interventions: Dietary Supplement: GLUCERNA SR®

INTERVENTIONS:
Dietary Supplement: SANZ®KINGWILL — 20g nutrition product (SANZ®KINGWILL) was used as extra meal at 10:00am and 15:00pm, respectively.
  Arms: Experimental group
Dietary Supplement: GLUCERNA SR® — 17.5g nutrition product (GLUCERNA SR®) was used as extra meal at 10:00am and 15:00pm, respectively.
  Arms: Control group

SUMMARY:
A prospective, multicenter, randomized controlled trial including about 60 Gestational Diabetes Mellitus patients (GDM) in Beijing will be included to evaluate the effectiveness and safety of nutrition product (SANZ®KINGWILL) in GDM patients, based on Continuous Glucose Monitoring (San MediTech CGM-303).

DETAILED DESCRIPTION:
This study will recruit pregnant women who were diagnosed as GDM by 75g Oral glucose tolerance test (OGTT) in 2nd trimester and followed up for 1month. A total of 60 GDM patients were expected to be enrolled. Using the double-blind method, they were randomly divided into two groups: experimental group and control group. Both of the two groups were provided medical nutrition treatment by nutritionist after GDM was diagnosed and CGM equipment (San MediTech CGM-303) was worn. Blood and urine samples were collected. At the following two days, oatmeal (SHIZHUANG) was used as extra meal at 10:00am and 15:00pm in both groups. In the next 4 weeks experimental group was provided with the domestic nutrition product (SANZ®KINGWILL), while existing products (GLUCERNA SR®) for control group as their extra meals at 10:00am and 15:00pm. In the last day, CGM equipment (San MediTech CGM-303) was removed and blood and urine samples were collected.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women aged 22 to 40 years old 2. Diagnosed as gestational diabetes mellitus 3. Signed informed consent

Exclusion Criteria:

* 1. GDM patient who is no longer suitable to continue pregnancy. 2. Patients who use any hypoglycemic drugs or any type of similar products. 3. Patients who have diseases severely affected the nutrition product digestion and absorption.

  4. Patients with severe heart, liver, kidney dysfunction, mental retardation, dyscrasia, etc.

  5. Patients who cannot tolerate enteral nutrition. 6. Patients with other conditions which investigator believes they are not eligible for this study.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Number of other product-related/possibly related adverse events or serious adverse events | 4 weeks
  Number of other product-related/possibly related adverse events or serious adverse events
Changes of Weight | 4 weeks
Area under the blood glucose curve (AUC) | 4 weeks
  Area under the blood glucose curve (AUC) by CGM within 2 hours of using the nutrition product.
Blood glucose control outcome | 4 weeks
  Fasting blood glucose
Glycated albumin level | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuli He, attending, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No